CLINICAL TRIAL: NCT00930605
Title: A Phase II Study of Alemtuzumab in Combination With CHOP and ESHAP as First-Line Treatment in Peripheral T-Cell Lymphoma
Brief Title: The Effectiveness of Alemtuzumab Given in Combination With CHOP and ESHAP in Patients Newly Diagnosed With Peripheral T-Cell Lymphoma (PTCL)
Acronym: C+CHOP/ESHAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Prof.Tanin Intragumtornchai, Division of Hematology and Stem Cell Transplant, Department of Medicine, Faculty of Medicine, Chulalongkorn University, King Chulalongkorn Memorial Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH011001
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — ESHAP regimen; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alemtuzumab combination with CHOP and ESHAP (Experimental): Alemtuzumab 30 mg/day is given subcutaneously on day 1-3 of cycle 1-5. CHOP alternate with ESHAP is given every 21 days for a total of 6 course.
  Interventions: Drug: CHOP regimen alternate with ESHAP regimen; Drug: Alemtuzumab

INTERVENTIONS:
Drug: CHOP regimen alternate with ESHAP regimen — CHOP alternate with ESHAP is given every 21 days for a total of 6 course.
Drug: Alemtuzumab — Alemtuzumab 30 mg/day is given subcutaneously on day 1-3 of cycle 1-5.

SUMMARY:
1. Primary Research Question What are the rates of complete response (CR), partial response (PR), progression free survival (PFS) and overall survival (OS) in adult patients newly diagnosed with Peripheral T-Cell Lymphoma (PTCL) who are treated with alemtuzumab given in combination with CHOP (cyclophosphamide, doxorubicin, vincristine and prednisolone) and ESHAP (etoposide, methylprednisolone, cisplatin, cytosine arabinoside) administered as an up-front treatment?
2. Secondary Research Question What is the incidence of life-threatening toxicities (grade 3 and 4, according to WHO criteria, Appendix A) in the patients?

DETAILED DESCRIPTION:
Alemtuzumab (Campath-1H) is a humanized monoclonal antibody that targets CD52, a cell surface protein present at high density on most normal and malignant B and T lymphocytes.

CHOP (cyclophosphamide, doxorubicin, vincristine and prednisolone) is currently regarded as a standard chemotherapy regimen for patients with newly diagnosed NHL.

ESHAP (etoposide, methylprednisolone, cisplatin, cytosine arabinoside) chemotherapy was invented in 1994. The regimen was aimed to salvage NHL patients who were relapsing or refractory to front-line, mostly doxorubicin-based, chemotherapy.Major toxicities were myelosuppression; 30% of the patients developed febrile neutropenia and was admitted for parenteral antibiotics. Treatment-related deaths, mostly from uncontrolled sepsis, occurred in 4% of the patients. Because of its efficacy and tolerable toxicities, at present, ESHAP is one of the salvage chemotherapy regimens most frequently administered to patients especially prior to autologous stem cell transplantation.

Recently, our unit had reported the efficacy of the combination of standard CHOP chemotherapy and ESHAP and high-dose therapy with autologous stem cell transplantation or rituximab given as upfront therapy in patients newly diagnosed as poor prognosis aggressive NHL (high- and high-intermediate risk groups according to the international index).15,16 According to the previous institutional experience as well as the efficacy of the combination of CHOP and ESHAP in patients with high-risk aggressive lymphoma, we would like therefore to determine the outcome of alemtuzumab given in combination with CHOP and ESHAP in patients newly diagnosed with PTCL, the effectiveness of which has not been known.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of one of the following histologic types according to the WHO classification:

   * Angioimmunoblastic T-cell lymphoma
   * Extranodal NK/T-cell lymphoma, nasal type
   * Enteropathy-type T-cell lymphoma
   * Hepatosplenic gamma-delta T-cell lymphoma
   * Subcutaneous panniculitis-like T-cell lymphoma
   * Anaplastic large-cell lymphoma, T/null cell, primary systemic type
   * Peripheral T-cell lymphoma, not otherwise characterized

     * All biopsy specimens including patients whose diagnosis have been made outside King Chulalongkorn Memorial Hospital will be reviewed by an expert hematopathologist at Department of Pathology, King Chulalongkorn Memorial Hospital.
2. Newly diagnosed, age 15 - 65 years.
3. Complete work up for baseline evaluation and measurement (Appendix B).
4. Patient's free written inform consent.

Exclusion Criteria:

1. Patients with a known hypersensitivity to murine proteins or to any component of alemtuzumab.
2. Patients who have received prior antilymphoma treatment with chemotherapy or radiotherapy.
3. Patients with poor performance status (PS; ECOG criteria of 3-4)(Appendix C).
4. Serologic evidence of human immunodeficiency virus exposure.
5. Patients with history of impaired cardiac status or myocardial infarction.
6. Patients with serum creatinine > 1.8 mg/dl, bilirubin > 1.5 times upper limit of normal range, SGOT or SGPT > 3 times upper limit of normal range, unless due to tumor involvement.
7. Patients with active uncontrolled infection, active non-malignant gastric or duodenal ulcer, uncontrolled diabetes mellitus or other severe medical conditions which would preclude aggressive cytotoxic chemotherapy.
8. Pregnant or lactating women.
9. Serious medical or psychiatric illness which prevent informed consent.
10. Patients who are likely to lost to follow up (e.g., unwilling or difficult to return, cannot be contacted).

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-01; Primary Completion 2006-11 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The response to treatment and the treatment-related toxicity. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tanin Intragumtornchai, M.D., Principal Investigator — Division of Hematology and Stem Cell Transplant, Department of Medicine, Faculty of Medicine, Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand